CLINICAL TRIAL: NCT01845389
Title: Comparative Study Between Continuous Epidural Anesthesia Using Standard Epidural Catheter And Continuous Spinal Anesthesia Using Wiley™ Spinal Catheter In Geriatric Patients Undergoing TURP
Brief Title: Comparative Study Between Continuous Epidural Anesthesia And Continuous Spinal Anesthesia Using Wiley™ Spinal Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theodor Bilharz Research Institute (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Yasser Mostafa Samhan, Prof Dr, Theodor Bilharz Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Anesth-2013
Record Dates: First submitted 2013-04-26; First posted 2013-05-03 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Anesthesia; Adverse Effect, Spinal and Epidural
Keywords: Anesthesia; Regional; Epidural; Continuous spinal; Wiley Catheter; Geriatric; TURP
MeSH Terms: interventions — Injections, Epidural

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epidural (Experimental): epidural anesthesia was administered via a 20-gauge epidural catheter threaded cephalad through an 18 gauge needle identified by the loss of resistance method to air. Bupivacaine 0.5% 5 ml every 5 minutes for T10 sensory level
  Interventions: Device: Epidural (B. Braun)
- Spinal (Active Comparator): An18-gauge Tuohy peel-away epidural sheath was introduced into the epidural space by using loss of resistance technique to air. Epidural introducer was removed leaving epidural sheath to be a pathway for Wiley spinal catheter. A flexible, convenience curve 27-gauge atraumatic pencil point tip spinal needle was introduced through the epidural sheath. After CSF flow was confirmed, a 23-gauge flexible cannula was threaded over the spinal needle. Peel-away epidural sheath was removed and flexible cannula was continually advanced over the spinal needle into the intrathecal space cephaled. Bupivacaine 0.5% 0.5 ml every 5 minutes for T10 sensory level.
  Interventions: Device: Spinal (Wiley Spinal Catheter)

INTERVENTIONS:
Device: Epidural (B. Braun) — 20-gauge epidural catheter threaded cephalad through an 18 gauge needle identified by the loss of resistance method to air.
  Other Names: B. Braun
  Arms: Epidural
Device: Spinal (Wiley Spinal Catheter) — The Wiley Spinal® is an innovative Flexible Cannula over Needle designed for convenient intrathecal access. After dural puncture is achieved, an immediate dural seal is created. The flexible cannula is advanced off the needle ensuring cephalad delivery of medication.
  Other Names: Wiley Spinal Catheter
  Arms: Spinal

SUMMARY:
Geriatric patients have a significantly higher incidence of morbidity and morality during surgery compared with younger age group. Transurethral resection of the prostate (TURP) is the gold standard treatment for elderly patients with bladder outlet obstruction. Thus Regional techniques may be better tolerated in the elderly patients undergoing TURP having the advantages of minimizing blood loss and thromboembolic events. The Wiley Spinal™ (Epimed; Johnstown, NY) catheter is an innovative flexible cannula over needle designed for convenient intrathecal access that reduces PDPH. We hypothesized that using less anesthetics during continuous spinal anesthesia with the Wiley spinal catheter would offer more hemodynamic stability with less side effects when compared with continuous epidural anesthesia in patients undergoing TURP

DETAILED DESCRIPTION:
Geriatric patients have a significantly higher incidence of morbidity and morality during surgery compared with younger age group as they commonly have respiratory, circulatory and renal problems [1]. Transurethral resection of the prostate (TURP) is the gold standard treatment for elderly patients with bladder outlet obstruction. TURP procedure has been associated with high morbidity rate including bleeding, TURP syndrome, bladder perforation, hypothermia and disseminated intravascular coagulation during intraoperative and early postoperative period. Therefore, it becomes very important to keep a stable anesthesia that minimizes these side effects. Detection of such complications is quite difficult under general anesthesia as compared to regional anesthesia. Thus Regional techniques may be better tolerated in the elderly patients undergoing TURP having the advantages of minimizing blood loss and thromboembolic events [2].

Subarachnoid single dose injection provides a potent blockade of fast onset while its extension and duration are difficult to predict [3]. Continuous epidural anesthesia with a catheter placement offers flexibility to extend, intensify, and maintain the block as well as providing postoperative analgesia [4]. Continuous spinal anesthesia consists of introducing a catheter in the subarachnoid space and maintaining blockade by repeated anesthetic injections. The possibility of fractionating local anesthetics dosage along time allows a fast onset with better blockade quality and less hemodynamic changes [5]. Recent study [6] reported that pain scores in patients received continuous spinal anesthesia were significantly lower than those received continuous femoral nerve block.

Advantages of continuous spinal anesthesia include the following: (a) Prior placement of the catheter in the induction area facilitates the surgical schedule. (b) Spinal anesthesia may be induced through the catheter after the patient has been positioned for surgery, thereby lessening the potential for hypotension. (c) The low doses of local anesthetic intermittently injected eliminate the possibility of systemic toxic reactions. (d) Repeated injection of small doses of local anesthetic solution facilitates obtaining the right level of anesthesia and decreases the cardiovascular instability during induction. (e) Employing a low dose of local anesthetic shortens the recovery period. (f) Anesthesia can be prolonged when the duration of surgery is uncertain. (g) A definite end point (aspiration of cerebrospinal fluid) assures that the catheter is in the right place and so enhances the likelihood of successful anesthesia. (h) Subarachnoid narcotics may be administered during a surgical procedure or continued into the recovery period to provide long-lasting postoperative analgesia [7].

The disadvantages of continuous spinal anesthesia are as follows: (a) Additional time is required to place the catheter in the right place, which may occasionally prove difficult. (b) Spinal headache is possible. (c) There is a potential for catheter breakage, infection, nerve trauma, and hemorrhage (these potential complications have, however, rarely been documented in previous clinical settings). The primary factor that has limited use of continuous spinal anesthesia is the belief that the large size of available spinal catheters requiring insertion through large spinal needles will result in an incidence of post dural puncture headache (PDPH) in young patients that is unacceptable [7].

The Wiley Spinal™ (Epimed; Johnstown, NY) catheter is an innovative flexible cannula over needle designed for convenient intrathecal access that reduces PDPH [8]. We hypothesized that using less anesthetics during continuous spinal anesthesia with the Wiley spinal catheter would offer more hemodynamic stability with less side effects when compared with continuous epidural anesthesia in patients undergoing TURP. The primary outcome of this study is the hemodynamic variability between both techniques. Secondary outcomes of interest are detection of adverse events including early and late neurological complications. Thus the aim of this prospective randomized study is to compare the efficacy of the continuous spinal anesthesia using the Wiley spinal catheter and continuous epidural anesthesia in geriatric patients undergoing TURP.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I, II or III
* geriatric male patients
* aged over 60 years
* scheduled for elective TURP under regional anesthesia

Exclusion Criteria:

* neurological diseases
* mental disturbance
* previous history of stroke
* severe cardiopulmonary disorders
* clinically significant coagulopathy
* lumbar disc herniation
* previous back surgery
* infection at the injection site
* body mass index greater than 35 kg/m2
* hypersensitivity to amide local anesthetics

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-06; Primary Completion 2013-09 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Mean arterial blood pressure | Participants will be followed for the duration of surgery, an expected average of 90 minutes
  Non- invasive blood pressure will be recorded before administering anesthesia, immediately after placing the catheter, every 1min for the first 10 min, then every 5 min till end of the operation.

SECONDARY OUTCOMES:
Heart rate | Participants will be followed for the duration of surgery, an expected average of 90 minutes
  Heart rate will be recorded before administering anesthesia, immediately after placing the catheter, every 1min for the first 10 min, then every 5 min till end of the operation.
detection of adverse events | 30 days
  failure of regional anesthesia (unilateral or patchy block), pruritus, dizziness, nausea, vomiting, itching, PDPH and symptoms suggestive of neurologic damage (back pain, numbness, weakness or pain in legs, and bladder or bowel dysfunction)
Characteristics of sensory block | Two minutes after injection of local anesthetic until resolution of the block (about 6 hours postoperatively)
  A pinprick test is recorded 2 minutes after local anesthetic injection the every 2 minutes for the first 15 minutes then every 10 minutes till the end of operation then every 30 minutes until resolution of the block.
Characteristics of motor block | Two minutes after injection of local anesthetic until resolution of the block (about 6 hours postoperatively)
  Modified Bromage scale is recorded 2 minutes after local anesthetic injection the every 2 minutes for the first 15 minutes then every 10 minutes till the end of operation then every 30 minutes until resolution of the block.
Time to first analgesic injection | Every hour postoperatively up to 10 hours.
  0-10 visual analogue scale (VAS) (0: no pain at all, 10: maximum imaginable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Reeham S Ebeid, MD, Principal Investigator — Theodor Bilharz Research Institute
Locations (2):
- Egypt (2):
  - Kasr El Aini University Hospital, Cairo
  - Theodor Bilharz Research Institute, Giza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kramer S, Wenk M, Fischer G, Mollmann M, Popping DM. Continuous spinal anesthesia versus continuous femoral nerve block for elective total knee replacement. Minerva Anestesiol. 2011 Apr;77(4):394-400. Epub 2011 Feb 1. PMID 21483383
- [Background] Ozmen S, Kosar A, Soyupek S, Armagan A, Hoscan MB, Aydin C. The selection of the regional anaesthesia in the transurethral resection of the prostate (TURP) operation. Int Urol Nephrol. 2003;35(4):507-12. doi: 10.1023/b:urol.0000025616.21293.6c. PMID 15198156
- [Background] Palmer CM. Continuous spinal anesthesia and analgesia in obstetrics. Anesth Analg. 2010 Dec;111(6):1476-9. doi: 10.1213/ANE.0b013e3181f7e3f4. Epub 2010 Oct 1. PMID 20889935
- [Background] Tao W, Nguyen AP, Ogunnaike BO, Craig MG. Use of a 23-gauge continuous spinal catheter for labor analgesia: a case series. Int J Obstet Anesth. 2011 Oct;20(4):351-4. doi: 10.1016/j.ijoa.2011.07.010. Epub 2011 Sep 9. PMID 21907561
- See also: Home page of Theodor Bilharz Research Institute — http://www.tbri.sci.eg